CLINICAL TRIAL: NCT05593770
Title: International Sites: CONNECTS Master Protocol for Clinical Trials Targeting Macro-, Micro-immuno-thrombosis, Vascular Hyperinflammation, and Hypercoagulability and Renin-angiotensin-aldosterone System (RAAS) in Hospitalized Patients With COVID-19 (ACTIV-4 Host Tissue)
Brief Title: International Sites: Novel Experimental COVID-19 Therapies Affecting Host Response
Acronym: NECTAR
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Following a meeting of the DSMB on 20th September 2023, the recommendation was made to the sponsor on 26th September 2023 that the Fostamatinib arm of the trial ceases enrolment and study medication is discontinued immediately.
Sponsor: NEAT ID Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTIV-4
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; SARS-CoV2 Infection; Coronavirus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — fostamatinib

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a two-step process: 1) The participant will first be randomized in an m:1 ratio to receive an active study drug or placebo, where m represents the number of study drug arms for which the participant is eligible. 2) The participant will then be randomly assigned with equal probability to one of the study drug arms. Participants will receive the corresponding study drug or matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Which study drug arm the participant enters will be known to the research sites and the participants, but assignment to active versus placebo will be blinded. The randomized assignment, concealed from the research team, will be transmitted to the site pharmacy, who will provide study medication. The participant, treating clinicians, study personnel (other than the unblinded statistician who will prepare closed DSMB interim reports), and outcome assessors will all remain blinded to group assignment until after the database is locked and blinded analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fostamatinib (Experimental): An investigational oral spleen tyrosine kinase inhibitor.
  Interventions: Drug: Fostamatinib
- Placebo (Placebo Comparator): Orange film-coated, plain, bioconvex tablets for fostamatinib.
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib100-150mg orally twice daily for 14 days or 28 doses. Study medication will be continued as an outpatient if the patient is discharged prior to completing 28 doses.
  Arms: Fostamatinib
Drug: Placebo — Orange film-coated, plain bioconvex tablets orally twice daily for 14 days or 28 doses for fostamatinib. Study medication will be continued as an outpatient if the patient is discharged prior to completing 28 doses.
  Arms: Placebo

SUMMARY:
The overarching goal of the Master Protocol is to find effective strategies for inpatient management of patients with COVID-19. Therapeutic goals for patients hospitalized for COVID-19 include hastening recovery and preventing progression to critical illness, multiorgan failure, or death. Our objective is to determine whether modulating the host tissue response improves clinical outcomes among patients with COVID-19.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which causes coronavirus disease 2019 (COVID-19), has resulted in a global pandemic. The clinical spectrum of COVID-19 infection is broad, encompassing asymptomatic infection, mild upper respiratory tract illness, and severe viral pneumonia with respiratory failure and death. Between 13 and 40% of patients become hospitalized, up to 30% of those hospitalized require admission for intensive care, and there is a 13% inpatient mortality rate. The reasons for hospitalization include respiratory support, as well as support for failure of other organs, including the heart and kidneys. The risk of thrombotic complications is increased, even when compared to other viral respiratory illnesses, such as influenza. While 82% of hospitalized patients with COVID-19 are ultimately discharged alive, median length of stay is 10-13 days.

Early work in treating COVID-19 has focused on preventing worsening of the initial clinical presentation to prevent hospitalization and disease progression to organ failure and death. Studies conducted under this Master Host Tissue Protocol are expected to extend our knowledge of how to manage patients who are hospitalized for COVID-19 illness. Our objective is to determine whether modulating the host tissue response improves clinical outcomes among patients with COVID-19. This Master Protocol is a randomized, placebo-controlled trial of agents targeting the host response in COVID-19 in hospitalized patients with hypoxemia. The Master Host Tissue Protocol is designed to be flexible in the number of study arms, the use of a single placebo group, and the stopping and adding of new therapies. Our primary outcome is oxygen free days through day 28. This is defined as days alive and without supplemental oxygen use during the first 28 days following randomization. Patients who die on or before day 28 are assigned -1 oxygen free days.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized for COVID-19
2. ≥18 years of age
3. SARS-CoV-2 infection, documented by:

   1. nucleic acid test (NAT) or equivalent testing within 3 days prior to randomization OR
   2. documented by NAT or equivalent testing more than 3 days prior to randomization AND progressive disease suggestive of ongoing SARS-CoV-2 infection per the responsible investigator (For non-NAT tests, only those deemed with equivalent specificity to NAT by the protocol team will be allowed. A central list of allowed non- NAT tests is maintained in Appendix E. Appendix E. Non-NAT Tests Deemed with Equivalent Specificity to NAT by the Protocol Team).
4. Hypoxemia, defined as SpO2 <92% on room air, new receipt of supplemental oxygen to maintain SpO2 ≥92%, or increased supplemental oxygen to maintain SpO2 ≥92% for a patient on chronic oxygen therapy
5. Symptoms or signs of acute COVID-19, defined as one or more of the following:

   1. cough
   2. reported or documented body temperature of 100.4 degrees Fahrenheit or greater
   3. shortness of breath
   4. chest pain
   5. infiltrates on chest imaging (x-ray, CT scan, lung ultrasound)

Exclusion Criteria:

1. Onset of COVID-19 symptom fulfilling inclusion criterion #5 >14 days prior to randomization
2. Hospitalized with hypoxemia (as defined in inclusion #4) for >72 hours prior to randomization (the 72-hour window for randomization begins when the patient first meets the hypoxemia inclusion criteria after hospital admission)
3. Pregnancy
4. Breastfeeding
5. Prisoners
6. End-stage renal disease (ESRD) on dialysis
7. Patient undergoing comfort care measures only such that treatment focuses on end-of- life symptom management over prolongation of life.
8. The treating clinician expects inability to participate in study procedures or participation would not be in the best interests of the patient
9. Known allergy/hypersensitivity to IMP or its excipients

Fostamatinib Arm-Specific Exclusion Criteria:

The following exclusion criteria differ from the master protocol criteria:

1. Randomized in another trial evaluating fostamatinib in the prior 30 days

Study arm exclusion criteria measured within 24 hours prior to randomization:

1. AST or ALT ≥ 5 × upper limit of normal (ULN) or ALT or AST ≥ 3 × ULN and total bilirubin ≥ 2 × ULN
2. SBP > 160 mmHg or DBP > 100 mmHg at the time of screening and randomization
3. ANC < 1000/mL
4. Patient is anticipated to require a strong CYP3A inhibitor (Atazanavir, Certinib, Clarithromycin, Cobicistat and cobicistat-containing coformulations, Idelalisib,Indinavir, Itraconazole, Ketoconazole, Levoketoconazole, Lonafarnib, Lopinavir, Mifeprostone, Mibefradil, Nefazodone, Nelfinavir, Ombitasvir-paritaprevir-ritonavir plus dasabuvir, Posaconazole, Ribociclib Ritonavir, Saquinavir, Telithromycin, Troleandomycin, Tucatinib, Voriconazole) from randomization to 21 days post-randomization. For a full list of CYP3A4 substrates, please reference this regularly updated list: https://drug-interactions.medicine.iu.edu/MainTable.aspx.
5. Patient unable to participate or declines participation in the fostamatinib arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Pozniak, Prof, Principal Investigator — NEAT ID
Locations (21):
- Brazil (3):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital Federal dos Servidores do Estado, Rio de Janeiro
  - Instituto Nacional de Infectologia Evandro Chagas, Rio de Janeiro
- Germany (2):
  - University Hospital Bonn, Bonn
  - University of Frankfurt, Frankfurt
- Italy (4):
  - Ente Ospedaliero Ospedali Galliera, Genova
  - San Paolo Hospital - ASST Santi Paolo e Carlo, Milan
  - San Raffaele Turro Hospital, Milan
  - University of Milan, Milan
- South Africa (3):
  - Worthwhile Clinical Trials (WWCT Lakeview Hospital), Benoni
  - Clinical HIV Research Unit - Helen Joseph Hospital (WITS CHRU), Johannesburg
  - Global Clinical Trials (Pty) Ltd, Pretoria
- Spain (9):
  - Hospital Clinic Barcelona, Barcelona, Villarroel
  - Hospital General Universitario de Elche, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Universidad de Valladolid - Hospital Universitario Río Hortega, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were over 18 years old with documented SARS-COV-2 infection confirmed by nucleic acid test. Participants were assigned to receive either the active Fostamatinib drug or matching placebo.
Groups:
- Placebo: Orange film-coated, plain, bioconvex tablets for fostamatinib.
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
  Placebo: Orange film-coated, plain bioconvex tablets orally twice daily for 14 days or 28 doses for fostamatinib. Study medication will be continued as an outpatient if the patient is discharged prior to completing 28 doses.
Period: Overall Study
Arm/Group | Fostamatinib | Placebo
Started | 14 | 14
Completed | 12 | 9
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Population: Participants were over 18 years old hospitalised with documented SARS-COV-2 infection confirmed by nucleic acid test. Participants were assigned to one either the Fostamatinib the active drug or matching placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 10 | 11 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Brazil | 1 | 0 | 1
  South Africa | 2 | 3 | 5
  Italy | 1 | 1 | 2
  Germany | 0 | 1 | 1
  Spain | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Free Days Through Day 28
Description: This is defined as days alive and without supplemental oxygen use during the first 28 days following randomization. Patients who die on or before day 28 are assigned -1 oxygen free days. Patients will be considered to be receiving supplemental oxygen therapy when they are receiving any of the following: supplemental oxygen by nasal cannula, supplemental oxygen by face mask, high flow nasal cannula (HFNC), non-invasive ventilation (NIV), invasive mechanical ventilation (IMV), or extracorporeal membrane oxygenation (ECMO).
Time Frame: Day 1 to Day 28
Population: The number of participants enrolled by international sites was insufficient for analysis due to the early termination of the trial. This analysis was performed on all participants enrolled to the fostamatinib arm of the ACTIV-4 Host Tissue platform (United states + International sites).The global fostamatinib arm of the ACTIV 4 study enrolled 400 participants, of which 28 were included from international sites and the results are reported in a separate Clinicaltrials.gov record, ref NCT04924660
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 199 | 201
days | 13.4 (12.4) | 14.2 (12.1)

2. Secondary Outcome: In-hospital Mortality
Description: Number of patients who die during hospitalization
Time Frame: Day 1 to hospital discharge or Day 90 whichever comes first
Population: Participants who lacked outcome data were not included in the analysis. Ineligible participants or those who didn't receive the treatment were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 1 | 1

3. Secondary Outcome: Alive and Oxygen Free at Day 14
Description: Number of patients oxygen free at day 14. Patients will be considered to be receiving supplemental oxygen therapy when they are receiving any of the following: supplemental oxygen by nasal cannula, supplemental oxygen by face mask, high flow nasal cannula (HFNC), non-invasive ventilation (NIV), invasive mechanical ventilation (IMV), or extracorporeal membrane oxygenation (ECMO).
Time Frame: Day 1 to Day 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 10 | 8

4. Secondary Outcome: Alive and Oxygen Free at Day 28
Description: Number of patients oxygen free at day 28. Patients will be considered to be receiving supplemental oxygen therapy when they are receiving any of the following: supplemental oxygen by nasal cannula, supplemental oxygen by face mask, high flow nasal cannula (HFNC), non-invasive ventilation (NIV), invasive mechanical ventilation (IMV), or extracorporeal membrane oxygenation (ECMO)
Time Frame: Day 1 to Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 11 | 9

5. Secondary Outcome: Alive and Free of New Invasive Mechanical Ventilation at Day 28
Description: Number of patients alive free of new invasive mechanical ventilation at day 28
Time Frame: Day 1 to Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 12 | 11

6. Secondary Outcome: 28-day Mortality
Description: Number of patients who have died at Day 28
Time Frame: Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 1 | 1

7. Secondary Outcome: 60-day Mortality
Description: Number of patients who have died at Day 60
Time Frame: Day 60
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 1 | 2

8. Secondary Outcome: 90-day Mortality
Description: Number of participants mortality at Day 90
Time Frame: Day 90
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 12 | 12
Participants | 1 | 3

9. Secondary Outcome: Clinical Status Assessed Using World Health Organization (WHO) 8-point Ordinal Scale at Day 14
Description: Number of participants who fell within the ordinal scale per the below criteria. A higher score indicates a worse outcome.
  1. Ambulatory - Not hospitalized and no limitation of activities
  2. Ambulatory - Not hospitalized with limitation of activities or home oxygen use
  3. Hospitalized Mild Disease - Hospitalized, no oxygen therapy
  4. Hospitalized Mild Disease - Hospitalized, oxygen by mask or nasal prongs
  5. Hospitalized Severe Disease - Non-invasive ventilation or high-flow nasal cannula
  6. Hospitalized Severe Disease -Invasive mechanical ventilation
  7. Hospitalized Severe Disease - Invasive mechanical ventilation plus additional organ support with- vasopressors, RRT, or ECMO
  8. Dead
Time Frame: Day 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
Participants
  Score 1 | 8 | 6
  Score 2 | 3 | 1
  Score 3 | 0 | 1
  Score 4 | 1 | 3
  Score 5 | 0 | 0
  Score 6 | 0 | 0
  Score 7 | 0 | 0
  Score 8 | 1 | 1

10. Secondary Outcome: Clinical Status Assessed Using WHO 8-point Ordinal Scale at Day 28
Description: The number of participants who fell within the ordinal scale per the below criteria. A higher score means a worse outcome
  1. Ambulatory - Not hospitalized and no limitation of activities
  2. Ambulatory - Not hospitalized with limitation of activities or home oxygen use
  3. Hospitalized Mild Disease - Hospitalized, no oxygen therapy
  4. Hospitalized Mild Disease - Hospitalized, oxygen by mask or nasal prongs
  5. Hospitalized Severe Disease - Non-invasive ventilation or high-flow nasal cannula
  6. Hospitalized Severe Disease -Invasive mechanical ventilation
  7. Hospitalized Severe Disease - Invasive mechanical ventilation plus additional organ support with- vasopressors, RRT, or ECMO
  8. Dead
Time Frame: Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
Participants
  Score 1 | 9 | 7
  Score 2 | 1 | 3
  Score 3 | 1 | 1
  Score 4 | 1 | 0
  Score 5 | 0 | 0
  Score 6 | 0 | 0
  Score 7 | 0 | 0
  Score 8 | 1 | 1

11. Secondary Outcome: Clinical Status Assessed Using WHO 8-point Ordinal Scale at Day 60
Description: Number of participants who fell within the ordinal scale per the below criteria. A higher score means a worse outcome
  1. Ambulatory - Not hospitalized and no limitation of activities
  2. Ambulatory - Not hospitalized with limitation of activities or home oxygen use
  3. Hospitalized Mild Disease - Hospitalized, no oxygen therapy
  4. Hospitalized Mild Disease - Hospitalized, oxygen by mask or nasal prongs
  5. Hospitalized Severe Disease - Non-invasive ventilation or high-flow nasal cannula
  6. Hospitalized Severe Disease -Invasive mechanical ventilation
  7. Hospitalized Severe Disease - Invasive mechanical ventilation plus additional organ support with- vasopressors, RRT, or ECMO
  8. Dead
Time Frame: Day 60
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 11 | 12
Participants
  Score 1 | 7 | 7
  Score 2 | 2 | 1
  Score 3 | 0 | 1
  Score 4 | 1 | 1
  Score 5 | 0 | 0
  Score 6 | 0 | 0
  Score 7 | 0 | 0
  Score 8 | 1 | 2

12. Secondary Outcome: Hospital-free Days Through Day 28
Description: Days alive and not hospitalized during the first 28 days following randomization. Patients who die on or before day 28 are assigned a value -1.
Time Frame: Day 1 to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
days
  Spain: number analyzed (Participants) | 9 | 9
  Spain | 21.3 (8.2) | 19.5 (12.5)
  Brazil: number analyzed (Participants) | 1 | 0
  Brazil | -1 (NA) — Unable to provide standard deviation as only 1 participant affected |
  Germany: number analyzed (Participants) | 0 | 1
  Germany |  | 0 (NA) — Unable to provide standard deviation as only 1 participant affected
  Italy: number analyzed (Participants) | 1 | 0
  Italy | 14 (NA) — Unable to provide standard deviation as only 1 participant affected |
  South Africa: number analyzed (Participants) | 2 | 2
  South Africa | 25.5 (3.5) | 26.5 (0.7)

13. Secondary Outcome: Ventilator-free Days Through Day 28
Description: Days alive and not receiving mechanical ventilation during the first 28 days following randomization. Patients who die on or before day 28 are assigned a value -1.
Time Frame: Day 1 to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
days
  Spain: number analyzed (Participants) | 9 | 9
  Spain | 21.3 (8.2) | 19.5 (12.5)
  Brazil: number analyzed (Participants) | 1 | 0
  Brazil | -1 (NA) — Unable to provide standard deviation as only 1 participant affected |
  Germany: number analyzed (Participants) | 0 | 1
  Germany |  | 0 (NA) — Unable to provide standard deviation as only 1 participant affected
  Italy: number analyzed (Participants) | 1 | 0
  Italy | 14 (NA) — Unable to provide standard deviation as only 1 participant affected |
  South Africa: number analyzed (Participants) | 2 | 2
  South Africa | 25.3 (3.5) | 26.5 (0.7)

14. Secondary Outcome: Respiratory Failure-free Days Through Day 28
Description: Days alive and not in respiratory failure during the first 28 days following randomization. A respiratory failure-free day is defined as a day alive without the use of HFNC, NIV, IMV, or (ECMO). Patients who die on or before day 28 are assigned a value -1.
Time Frame: Day 1 to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 13 | 12
days
  Spain: number analyzed (Participants) | 9 | 9
  Spain | 21.3 (8.2) | 19.5 (12.5)
  Brazil: number analyzed (Participants) | 1 | 0
  Brazil | -1 (NA) — Unable to provide standard deviation as only 1 participant affected |
  Germany: number analyzed (Participants) | 0 | 1
  Germany |  | 0 (NA) — Unable to provide standard deviation as only 1 participant affected
  Italy: number analyzed (Participants) | 1 | 0
  Italy | 14 (NA) — Unable to provide standard deviation as only 1 participant affected |
  South Africa: number analyzed (Participants) | 2 | 2
  South Africa | 25.3 (3.5) | 26.5 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from day 0-60, Mortality will be collected from day 0-90
Arm/Group | Fostamatinib | Placebo
All-Cause Mortality (participants affected / at risk) | 1/14 | 3/14
Serious Adverse Events (participants affected / at risk) | 8/14 | 5/14
Other Adverse Events (participants affected / at risk) | 8/14 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib (N=14) | Placebo (N=14)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib (N=14) | Placebo (N=14)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1)
Injection site phlebitis (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to DSMB findings of extremely low likelihood of the intervention having a beneficial effect on the primary outcome led to a small number of participants enrolled by international sites and analysis being performed with data from all participants (International and US sites) in the fostamatinib arm of the ACTIV-4 Host Tissue study. Results for all participants in the fostamatinib arm of the ACTIV-4 Host Tissue study are recorded in Clinicaltrials.gov record NCT04924660.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT05593770/Prot_SAP_000.pdf